CLINICAL TRIAL: NCT06854705
Title: Remodeling Maternal Health Care: Evaluating the Impact of Implementing the Midwifery Model of Care on Maternal and Neonatal Health Outcomes in Ethiopia (MiMoC Project)
Brief Title: Impact of Implementing the Midwifery Model of Care on Maternal and Neonatal Health Outcomes in Ethiopia
Acronym: MiMoC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debre Berhan University (Other)
Collaborators: Dalarna University (Other); Sophiahemmet University (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Solomon Hailemeskel Beshah, PhD, Debre Berhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DebreBerhanU; INV-075963 (Other Grant/Funding Number: Bill and Melinda Gets Foundation)
Record Dates: First submitted 2025-02-19; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Midwifery Continuity of Care Model; Maternal Health Outcomes; Neonatal Health Outcomes; Cost Effectiveness

STUDY DESIGN:
Intervention Model Description: The intervention group will receive a continuity of midwifery care model organized by a team of qualified midwives. In this model, antenatal, intrapartum, and postnatal care will be provided by a named (or primary) midwife, who works within a small team (4-8) of CoMC midwives to their cohort of women and will refer or consult an obstetrician in case of complications that requires specialized care. Each named midwife will be backed up by a partner midwife and other team colleagues. The CoMC team comprises 8 whole-time equivalent midwives, including an experienced senior midwife, who leads the team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiMoC Arm (intervention Group) (Experimental): the MiMoC Arm which will be the intervention group, will provide the continuity of midwifery care (CoMC) starting from antenatal care up to the postnatal period.
  Interventions: Other: Continuity of Midwifery care model
- standard care model (control group) (Active Comparator): Pregnant women who receive antenatal, intrapartum, and postnatal care following standard practice in Ethiopia will be assigned to the control group. An established practice followed the shared model of care in which responsibility is shared among different staff members, including midwives, nurses, health officers, and medical doctors.
  Interventions: Other: Standard care model

INTERVENTIONS:
Other: Continuity of Midwifery care model — The intervention group will receive a continuity of midwifery care model organized by a team of qualified midwives. In this model, antenatal, intrapartum, and postnatal care will be provided by a named (or primary) midwife, who works within a small team (4-8) of CoMC midwives to their cohort of women and will refer or consult an obstetrician in case of complications that requires specialized care. Each named midwife will be backed up by a partner midwife and other team colleagues. The CoMC team comprises 8 whole-time equivalent midwives, including an experienced senior midwife, who leads the team. Following a training needs assessment by the team leader, midwives will receive specialist training, provided by a team of clinical experts and educators, on how to work in midwife continuity models. Pregnant women receive their entire antenatal, intrapartum, and postnatal care from one of the participating CoMC midwives.
  Arms: MiMoC Arm (intervention Group)
Other: Standard care model — Pregnant women who receive antenatal, intrapartum, and postnatal care following standard practice in Ethiopia will be assigned to the control group. An established practice followed the shared model of care in which responsibility is shared among different staff members, including midwives, nurses, health officers, and medical doctors. Midwives and other health care providers worked conventional eight-hour shifts and handed over care to the next health care provider coming on duty during the next shift. In this model of care, each unit of care had its staff working independently. Besides, the health care provider assigned to the postnatal ward will be responsible for immediate postnatal care. After discharge, each woman in this group become the responsibility of a different group of healthcare providers (usually midwives or nurses) in the family planning and immunization room.
  Arms: standard care model (control group)

SUMMARY:
Background: The Continuity of Midwifery Care (CoMC) is a maternity care model used in some high-income countries. In this model, a dedicated group of midwives supports women throughout pregnancy, labor, and the early postnatal period. This model has been shown to improve maternal and neonatal outcomes and enhance maternal satisfaction. However, its effectiveness in low-and middle-income countries remains uncertain.

Purpose and Aim of the Study: This study aims to evaluate whether CoMC, supported by midwife-led birthing centers, improves maternal and neonatal health outcomes compared to the standard care model in Ethiopia.

Research Question: Does the CoMC model, integrated with midwife-led birthing centers, enhance maternal and neonatal outcomes compared to the standard maternal health care model? Additionally, does its implementation strengthen midwives' capacity to deliver quality care and increase the uptake of evidence-based practices in Ethiopia? Methods: A hybrid implementation-effectiveness, randomized, controlled, unblinded, parallel-group pilot trial will be conducted. The type 2 hybrid design will equally emphasize effectiveness and implementation outcomes. The study will take place in four randomly selected hospitals in the North Shoa Zone, Amhara regional state, Ethiopia, involving 1,654 pregnant women (<20 weeks gestation at first ANC visit). Participants will be randomly assigned to CoMC (Group A) or standard care (Group B) using a computer-generated scheme. Midwives will be organized into teams following the CoMC model. Women will receive study information during ANC visits and, if interested, will discuss participation with the CoMC team leader. Upon consent, they will be randomly allocated using a secure computerized system.

In the CoMC arm, women will receive care from a single midwife or a backup midwife throughout pregnancy, labor, birth, and the immediate postnatal period. In the standard care arm, multiple staff members will provide care at different times.

Outcomes: The primary maternal outcome is the proportion of women achieving spontaneous vaginal birth. The primary neonatal outcome is the proportion of neonates experiencing preterm birth. These outcomes will be analyzed using bivariable and multivariable generalized linear models (GLMs) with 95% confidence intervals.

DETAILED DESCRIPTION:
Background The World Health Organization (WHO) published a position paper in 2024 stating that Continuity of Midwifery Care (CoMC) models may improve maternal and child health by enabling women to develop relationships with the same caregivers throughout pregnancy, birth, and the postnatal period (1). Women receive care from a named midwife and a backup midwife from the same team, whom they have met before and feel familiar with. This close relationship helps women feel supported by a healthcare provider who knows their medical history and will care for them during labor, birth, and postpartum.

Traditionally, maternity care in Ethiopia has been fragmented, resembling a shared model of care where different healthcare providers assume midwifery roles at various stages. Women may not know their care providers or have previously met the professionals attending their labor. The research team behind this proposal has conducted several studies within the field. A quasi-experimental study among 1,178 low-risk pregnant mothers in four randomly selected primary hospitals in the North Shoa Zone, Amhara Region, demonstrated the successful implementation of a midwife continuity of care model (2). This study highlighted its potential to improve maternal and neonatal health outcomes, increase maternal satisfaction, enhance antenatal and postnatal care utilization, and save lives.

The purpose of this proposal is to increase evidence-based midwife-led practices and strengthen midwives' capacity to lead quality improvement initiatives in maternal and newborn health. The primary goal is to evaluate whether the Midwifery Model of Care (MiMoC), supported by midwife-led birthing centers, is more effective in improving maternal and neonatal health outcomes than the standard care model in Ethiopia. The study will also assess whether this continuous quality improvement initiative increases the uptake of evidence-based practices and enhances midwives' leadership in quality care.

Objectives

* Assess the impact of MiMoC, incorporating midwife-led birthing centers, on maternal health outcomes compared to the standard model of care.
* Evaluate the impact of MiMoC on neonatal health outcomes.
* Explore the experiences and perspectives of healthcare providers, mothers, and companions regarding the continuity of midwifery-led care.
* Measure the effect of MiMoC on the utilization of evidence-based midwife-led practices in health facilities.
* Assess midwives' capacity to lead quality improvement initiatives in a CoMC context.
* Evaluate the cost-effectiveness of MiMoC integrated with midwife-led birthing centers compared to the current maternal healthcare model.

Methods Between February 24, 2025, and February 23, 2026, 1,654 pregnant women in Debre Berhan with gestational ages of less than 24 weeks will be randomly allocated to receive either the MiMoC intervention or standard care. Randomization will occur at selected health facilities using a secure computerized system (MedSciNet). Effect-modifying and confounding factors will be considered in the analysis. Primary and secondary endpoints will be analyzed according to the intention-to-treat principle. Ethical approval has been obtained from the Swedish Ethical Review Board and the study is registered with ClinicalTrials.gov.

Study Design A hybrid implementation-effectiveness randomized controlled, unblinded, parallel-group pilot trial design will be used. A type 2 hybrid design will allow for equal focus on intervention effectiveness and implementation. A quality improvement approach will guide intervention implementation, and results will be reported following Consolidated Standards of Reporting Trials (CONSORT) guidelines.

Sample Size Estimation Sample size was determined using STATA software, based on prior research comparing maternal and neonatal outcomes in CoMC versus standard care in North Shoa Zone. The largest required sample size was based on the proportion of perineal tears (1.2% in CoMC vs. 3.6% in standard care), with a 95% confidence level and 80% power. Assuming a 15% loss to follow-up, 1,654 participants (827 per group) are required.

Randomization Process Eligible pregnant women receiving antenatal care at selected health facilities will be informed about the study and referred to the MiMoC team leader if interested. After providing written informed consent, participants will be randomized 1:1 into either the MiMoC or standard care group using a secure computerized system.

Implementation MiMoC, supported by midwife-led birthing centers, will be coordinated by Debre Berhan University Hakim Gizaw Teaching Hospital in collaboration with midwifery, obstetrics, gynecology, and pediatric departments. Investigators from Debre Berhan University and Sophiahemmet University (Sweden) will provide training on organizing and implementing MiMoC. Additional training for facility staff will be documented and evaluated. Biweekly digital meetings will support champions leading MiMoC implementation, using run charts to monitor key performance indicators.

Fidelity of Intervention Delivery Treatment fidelity will be monitored throughout training and intervention delivery. Midwives in the intervention group will be trained to adhere to clinical guidelines and maintain continuity of care. Fidelity will be assessed through midwife interviews, research team meetings, and medical record reviews. Measures include antenatal care completion, care continuity, referrals, and women's perceptions of provider continuity.

Outcome Variables

Maternal:

• Mode of birth, episiotomy, perineal trauma, labor augmentation, hemorrhage, prolonged/obstructed labor, maternal death (within 42 days), satisfaction with care, and healthcare utilization.

Neonatal:

• Birth status, perinatal death, APGAR scores, birth complications, birth weight, NICU admission, and early breastfeeding initiation.

Cost:

• Healthcare provider costs, including salaries, goods and services, and repair/maintenance costs, will be analyzed for cost-effectiveness.

Feasibility:

• Recruitment, attrition rates, fidelity (proportion of births attended by a known midwife), and clinical decision-making processes will be assessed.

Data Collection Independent data collection teams will be established in each hospital. Research assistants will ensure quality control in data collection and transfer to the central research center (Debre Berhan University and Sweden). Clinical data will be anonymized, with unique identification numbers assigned. Data collection will focus on maternal and neonatal health outcomes, adherence to MiMoC, and midwives' leadership in quality improvement.

Data Analysis

Intention-to-treat analysis will be used. Binary correlated data will be analyzed using McNemar's test, and differences between health facilities will be assessed using logistic regression. Training scores will be analyzed longitudinally using mixed model effects. Cost-effectiveness analysis will compare incremental costs and health outcomes, using the Incremental Cost-Effectiveness Ratio (ICER):

ICER = (Cost of MiMoC - Cost of Standard Care) / (Effect of MiMoC - Effect of Standard Care) Costs per patient will be estimated based on real-life healthcare use over pregnancy, labor, and the postnatal period.

Dissemination and Impact This research will generate evidence-based recommendations for scaling up MiMoC, supported by midwife-led birthing centers, to improve maternal and neonatal health outcomes in Ethiopia. The project aligns with Sustainable Development Goals 3 and 5, aiming to empower women and reduce maternal and neonatal mortality. Results will be disseminated to policymakers, healthcare providers, and communities through national and international conferences and peer-reviewed publications. If effective, MiMoC will be scaled to other regions and low- and middle-income countries. Policy briefs and implementation guidelines will be developed, and midwifery birthing centers will be established.

Ethical Considerations Ethical approval has been obtained from Debre Berhan University's Institutional Review Board and the Swedish National Ethical Review Board. The study will adhere to ethical research standards, including informed consent, data protection, inclusivity, and participant well-being.

ELIGIBILITY:
Inclusion Criteria:

* All sampled pregnant women above 18 years with gestational age less than 24 whole weeks at the first ANC booking at the Government Hospitals
* Singleton pregnancy, and
* low obstetric risk.

Exclusion Criteria:

* Women who plan to have an elective cesarean section or
* Women who have a history of medical or obstetric complications.
* pregnant women who are unable to provide valid information due to mental, hearing, speech, or other medical issues that could worsen their current pregnancy will also be excluded.
* pregnant mothers who are temporary residents and are expected to leave the study area before the 42-day postpartum period.
* Women with a history of medical and obstetrics complications.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1654 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Vaginal Birth | 12 months
  Proportion of women having a spontaneous vaginal birth.
preterm birth | 12 months
  The proportion of neonates who had a preterm birth.

REFERENCES:
- [Background] Hailemeskel S, Alemu K, Christensson K, Tesfahun E, Lindgren H. Midwife-led continuity of care improved maternal and neonatal health outcomes in north Shoa zone, Amhara regional state, Ethiopia: A quasi-experimental study. Women Birth. 2022 Jul;35(4):340-348. doi: 10.1016/j.wombi.2021.08.008. Epub 2021 Sep 3. PMID 34489211
- [Background] Transitioning to midwifery models of care: global position paper. Geneva: World Health Organization; 2024. Licence: CC BY-NC-SA 3.0 IGO.